CLINICAL TRIAL: NCT03827681
Title: A Randomised Controlled Trial to Study the Efficacy and Safety of TIPS (Trans Intrahepatic Portosystemic Shunt) Versus Self Expanding Metallic Stent (SEMS) in the Management of Refractory Variceal Bleed in Cirrhotics.
Brief Title: To Study the Efficacy and Safety of TIPS (Trans Intrahepatic Portosystemic Shunt) Versus Self Expanding Metallic Stent (SEMS) in the Management of Refractory Variceal Bleed in Cirrhotics.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-20
Record Dates: First submitted 2019-01-31; First posted 2019-02-01 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Liver Cirrhoses
MeSH Terms: interventions — Vasoconstrictor Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TIPS + Vasoactive Drug (Experimental)
  Interventions: Procedure: Trans Intrahepatic Portosystemic Shunt; Drug: Vasoactive Agent
- SEMS + Vasoactive Drug (Active Comparator)
  Interventions: Procedure: Self Expanding Metallic Stent; Drug: Vasoactive Agent

INTERVENTIONS:
Procedure: Trans Intrahepatic Portosystemic Shunt — * The most common approach is through the right internal jugular approach.
  * After infiltrating the puncture site with 2% lignocaine and puncturing the vein a guide wire is advanced into the IVC followed by a 9F/10F vascular sheath.
  * A wedged venogram is performed with a peripherally placed hepatic vein catheter, which may identify a portion of the portal vein to facilitate subsequent puncture.'
  * A stiff guide wire is then passed through the catheter and the vascular sheath is advanced into the right hepatic vein. With the vascular sheath in place a rigid needle with 15-20 degrees of distal angulation is advanced over the guide wire and through the vascular sheath to enter the hepatic vein.
  Arms: TIPS + Vasoactive Drug
Procedure: Self Expanding Metallic Stent — * At upper endoscopy, a 0.35 Superstiff radiological guidewire with a soft tip (supplied with the stent insertion kit) is delivered into the stomach under direct vision and the endoscope is removed.
  * The stent delivery device is then advanced over the guidewire into the stomach, and the distal portion of the stent delivery system is withdrawn to allow inflation of the gastric balloon.
  * The gastric balloon is then inflated with 100 mL of air, and the whole delivery system is withdrawn until resistance is felt, which signifies that the balloon is impacting at the cardia, thus anchoring the distal end of the stent during deployment.
  * After stent deployment, the gastric balloon is deflated and the stent delivery system is withdrawn. The stent is then examined endoscopically. When deployed, the stent is 135 mm long and 25 mm wide.
  Arms: SEMS + Vasoactive Drug
Drug: Vasoactive Agent — Vasoactive Agent

SUMMARY:
A total of 50 patients will be enrolled and will be randomized into either Group A(TIPS) or Group B (SEMS).

Primary end point of the study will be to compare efficacy of TIPS versus SEMS for survival at 6 week or Early re Bleed. All enrolled patients will also undergo HVPG measurement at baseline to stratify risk of failure to control bleed or early re-bleed.

Patient will be monitored for 5 days for re bleed, complications of therapy, worsening of Liver function tests and scores and efficacy of either treatment modality over other. Patient will be followed for 6 weeks to see for the primary end point.

ELIGIBILITY:
Inclusion Criteria:

- Consecutive patients of cirrhosis aged 18-70 years presenting with acute variceal Bleeding, who on endoscopy fail to control bleed or rebleeds within 5 days will be randomized.

Exclusion Criteria:

* Bleeding from non-variceal source
* Coagulopathy related bleed
* Bleeding from Gastric varices
* Any malignancy including HCC
* Main Portal vein thrombosis
* Patients in refractory shock
* Patients with severe cardiopulmonary disease
* Grade 4 Hepatic encephalopathy
* MELD > 25
* Multiorgan failure
* Active sepsis
* Pregnancy
* Failure to give consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-02-06 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Survival in both groups | 6 weeks

SECONDARY OUTCOMES:
Re-bleeding in both groups for 5 days from end of therapy | 5 days
Rebleeding in both groups | 6 weeks
Decompensation in both groups in the form of ascites or Hepatic Encephalopathy | 6 weeks
Adverse events in both groups | 6 weeks
Worsening of liver severity score in both groups. | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Singh S, Arora V, Maiwall R, Mukund A, Jindal A, Choudhry A, Kumar G, Sarin SK. TIPS Is Superior to SEMS in the Management of Refractory VARICEAL Bleed in Advanced Cirrhosis Patients (TIPSEMS-VB Trial). Liver Int. 2025 Aug;45(8):e70178. doi: 10.1111/liv.70178. PMID 40631454